CLINICAL TRIAL: NCT07303621
Title: Population Pharmacokinetics of Elexacaftor-tezacaftor-ivacaftor in a Paediatric Population
Acronym: IMPROVED
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0708; 2025-A01805-44 (Other: N° ID-RCB)
Record Dates: First submitted 2025-11-19; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Trikafta; Elexacaftor; Ivacaftor; Cystic Fibrosis; pharmacokinetics
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trikafta, Elexacaftor, Ivacaftor, Tezacaftor, Cystic Fibrosis, Population pharmacokinetics
  Interventions: Other: There is no intervention as this is a prospective pharmacokinetics study.

INTERVENTIONS:
Other: There is no intervention as this is a prospective pharmacokinetics study. — There is no intervention as this is a prospective pharmacokinetics study.

SUMMARY:
Cystic fibrosis is a rare, progressive genetic disease caused by a mutation in the CFTR (cystic fibrosis transmembrane conductance regulator) gene. Respiratory and nutritional effects are crucial to patients' prognosis. Since the early years of 2010, etiological treatment has been based on the use of CFTRm (CFTR modulator), which aim to restore the function of the mutated protein. Initially used as monotherapy and targeting a limited number of patients, CFTRm has gradually been extended to a larger number of patients, to the point where it now concerns 9 out of 10 patients, through the use of triple therapy with Elexacaftor-Tezacaftor-Ivacaftro (ETI) or Kaftrio(R).

The efficacy of triple therapy is spectacular, revolutionizing the prognosis of the disease. However, the potential for neuropsychological side-effects (20-50% depending on age, but more frequent in young children under 5) and hepatic side-effects (hepatic cytolysis) must be taken into account. A better understanding of pharmacokinetic variability in children, as well as the relationship between exposure to therapeutic effects and adverse reactions, is therefore particularly important.

The aim of this study is to measure the association between the pharmacokinetic parameters of Elexacaftor, Tezacaftor and Ivacaftor (plasma clearance and volume of distribution) and therapeutic or adverse effects in pediatric patients with cystic fibrosis treated with the combination.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 17 years old
* Having Cystic Fibrosis
* Treated by Elexacaftor/Tezacaftor and Ivacaftor (Trikafta® or Kaftrio®)

Exclusion Criteria:

* Allergy to previous CFTR modulator association (Ivacaftor, lumacaftor)
* Pregnant women
* Patient already enrolled in another study with CYP3A4 inhibitor
* Pulmonary transplant recipient

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population is from a tertiary care hospital. Children enrolled in the study are followed in the referral center for pediatric cystic fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Trough Concentration [Cmin] of Elexacaftor, Ivacaftor and Tezacaftor | 5 minutes pre-dosing 3 to 4 hours post-dosing 6 to 7 hours post-dosing
  Measure residual concentration of Elexacaftor, Ivacaftor and Tezacaftor
Maximum Plasma Concentration [Cmax] | 5 minutes pre-dosing 3 to 4 hours post-dosing 6 to 7 hours post-dosing
  Measured Cmax of Elexacaftor, Ivacaftor and Tezacaftor
Area Under the Concentration Time Curve between two administrations of Elexacaftor, Ivacaftor and Tezacaftor | 5 minutes pre-dosing 3 to 4 hours post-dosing 6 to 7 hours post-dosing
  Area under the concentration time curve between two administrations of (AUC0-tz) of Elexacaftor, Ivacaftor and Tezacaftor

SECONDARY OUTCOMES:
Number (Proportion) of Subjects with adverse events | 5 minutes pre-dosing 3 to 4 hours post-dosing 6 to 7 hours post-dosing
  Specific drug related adverse events such as hepatic impairment or neurocomportmental disorder will be monitored.
  All safety data will be analysed using descriptive statistics. Pharmacokinetics analysis will be used to monitor existing relationship between elexacaftor/tezacaftor and ivacaftor
Relationship between Pharmacokinetics and Cystic Fibrosis mutational status and Adverse Event | 5 minutes pre-dosing 3 to 4 hours post-dosing 6 to 7 hours post-dosing
Relationship between Pharmacokinetics/Toxixodynamic and Cystic Fibrosis mutational status | 5 minutes pre-dosing 3 to 4 hours post-dosing 6 to 7 hours post-dosing
Number of Participants with Clinically Significant Changes in Clinical Laboratory Evaluations | 5 minutes pre-dosing 3 to 4 hours post-dosing 6 to 7 hours post-dosing
  Area Under the Effect Time curve (AUEC) of Lung Clearance Index 2.5
Area Under the Effect Time curve (AUEC) of Sweat Chloride | 5 minutes pre-dosing 3 to 4 hours post-dosing 6 to 7 hours post-dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant (HFME), Bron, France